CLINICAL TRIAL: NCT04555070
Title: Assessment of The Direction and Severity of Root Canal Curvatures of the Permanent Mandibular First and Second Molars in a Sample of Egyptian Population Using CBCT: A Cross-Sectional Study
Brief Title: Assessment of Root Canal Curvatures of the Permanent Mandibular First and Second Molars in a Sample of Egyptian Population Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farid Medhat, principal investigator, Cairo University
Other Study IDs: ORAD7:1:1
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Prevalence of Curvatures in Root Canals; Direction of Curvatures in Root Canals; Severity of Curvatures in Root Canals
Keywords: Mandibular molars; Root canal curvature; Root canal complexity; CBCT

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study to assess variations in root canal curvatures of the Permanent Mandibular First and Second Molars in a Sample of Egyptian Population using cone beam computed tomography through retrospective data analysis

DETAILED DESCRIPTION:
A) Study design and setting

* Study Design: An observational Cross-sectional Study
* Setting and Location: Being a retrospective study, CBCT scans of Egyptian patients who have already been subjected to CBCT examination as part of their dental diagnosis and/or treatment planning will be included. The CBCT scans will be obtained from the data base available at the department of Oral and Maxillo-facial Radiology, Faculty of Dentistry, Cairo University, and a private Oral Radiology center, Cairo, Egypt.

B) Participants:

Based on sample size calculation, a sample of 272 canals of mandibular first and second permanent molars belonging to Egyptian individuals will be examined. The selection of the scans to be included will be based on the following eligibility criteria.

C) Variables:

* Details about variable

  1. Mesio-distal direction of root canal curvatures in the sagittal cuts.
  2. Bucco-lingual direction of root canal curvatures in the coronal cuts.
  3. Schneider's angle of root canals curvatures present in both coronal and sagittal cuts.

     D) Data Sources / Measurements:
     * Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.
     * Exposure parameters of the scans were varied depending on the individual patient's sizes.
     * CBCT scans showing mandibular first and second permanent molars with maximum 0.2 voxel sizes will be reviewed.
     * CBCT images will be analysed using Planmeca Romexis Viewer software, CBCT images will be analyzed in 2 planes; the root canal curvatures in the mesio-distal dimension from the sagittal section and the curvatures in the bucco-lingual dimension from the coronal sections, determining the direction of root canal curvatures.
     * For each image of canal trajectory, the number of curvatures and their angle will be recorded using Schneider's criteria (Schneider 1971) as follows; (5 degrees or less); as straight canal (10 to 20 degrees); as moderate curvature (25 to 70 degrees); as severe curvature
     * If the trajectory of the canal contained more than one curve, the additional curvatures were measured as described by Cunningham & Senia (1992) who measured Schneider's angle for each curve.
     * All CBCT scans will be interpreted by the main investigator, and 30% of the scans will be re-viewed by the same radiologist to assess intra-observer reliability with at least 2 weeks interval and by another experienced radiologist (co-supervisor) to assess inter-observer reliability.

     E) Addressing potential sources of bias:

     No source of bias. CBCT scans will be coded and interpreted by two oral and maxillofacial radiologists blinded from demographic data of the patients and from the results of each other.

     F) Study Size:

     This power analysis used percentage of curved canals at the cervical third in sagittal plane as the primary outcome. Based upon the results of Estrela C et al (2015), the percentage was 77%. Using alpha (α) level of (5%), acceptable margin of error = 5%; the minimum estimated sample size was 272 canals. Sample size calculation was performed using Epi Info 7.2.2.2.

     G) Sampling strategy: The sample will be collected by simple random sampling. H) Quantitative variables
* Handling of quantitative variables in analyses The number of root canals of permanent mandibular first and second molars of Egyptian individuals with root canal curvatures will be counted to estimate the variations in the Egyptian population.

Severity of curvatures will be estimated using Schneider's method. The direction of curvatures will be detected from sagittal and coronal cuts.

I) Statistical methods:

*Statistical methods. Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Scienceaszxs), version 21 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans should show

  * Fully maturated and erupted mandibular permanent first and second molars of Egyptian patients above 16 years old.
  * Intact molars' roots without fractures or cracks.
  * Mandibular permanent first and second molars without posts or previous root canal treatment.
  * Full extension of mandibular first and second molars using different fields of view and maximum 0.2 mm voxel resolution will be included

Exclusion Criteria:

* • Evidence of apicectomy or peri-apical surgery.

  * Mandibular molars with developmental anomalies.
  * External or Internal Root resorption.
  * Root Canal Calcification.
  * Previous Root Canal treatment or posts.
  * Presence of Root caries.
  * Tomographic images of poor quality or artifacts interfering with the detection of root canals.

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
prevalence of root canal curvatures in cervical third of roots in mandibular first and second molars | one year

SECONDARY OUTCOMES:
prevalence of root canal curvatures in middle third of roots in mandibular first and second molars | one year

OTHER OUTCOMES:
prevalence of root canal curvatures in apival third of roots in mandibular first and second molars | one year
severity of root canal curvatures using Schneider's method | one year
direction of root canal curvatures | one year